CLINICAL TRIAL: NCT05669469
Title: Upper Airway of Women With Obstructive Sleep Apnea Changes After Bariatric Surgery and a Possible Influence of Menopause
Brief Title: Upper Airway of Women With Obstructive Sleep Apnea After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Michel Burihan Cahali (Other)
Collaborators: Carolina Ferraz de Paula Soares (Unknown)
Responsible Party: Sponsor-Investigator, Michel Burihan Cahali, Postgraduate supervisor and collaborating professor of Otorhinolaryngology at FMUSP, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Other Study IDs: 66609117.9.0000.0065
Record Dates: First submitted 2022-11-12; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Sleep Apnea; Obesity
Keywords: Sleep Apnea; Obesity; Bariatric Surgery
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — 1) gastric pouch creation, 2) creation of biliopancreatic limb, 3) jejunojejunostomy creation, and 4) creation of gastrojejunostomy.
  Other Names: surgical weight loss; Y-Roux

SUMMARY:
Evaluation of upper airway with Magnetic Resonance and polysomnographic at the pre and post operative of 23 women having undergone bariatric surgery (with the Y-Roux technique) for treatment of obesity.

DETAILED DESCRIPTION:
The the present study aims at describing the modifications occurring in the upper airway (UA) and the impact of such modifications on the severity of obstructive sleep apnea after bariatric surgery in women who have obstructive sleep apnea (OSA). The hypothesis is that the massive weight loss after bariatric surgery on OSA women could modify the UA more intensely than previously reported by other therapies for weight loss and that the menopause status may influence the likely reshaping of UA after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with a recommendation and considered apt for bariatric surgery by the multi-professional group
* aged between 18 and 70
* with a residual (after the 16-week period) BMI above 35 kg/m2
* polysomnographic obstructive sleep apnea diagnosis: Apnea-Hypopnea Index (AHI) above 5 events per hour associated with a co-morbidity and/or complaints of snoring.

Exclusion Criteria:

* patients with body weight above 180 kg - for the impossibility of having a magnetic resonance (MR)
* carrying metal artifacts which contraindicate the performing of MR
* patients with a history of pharyngeal or neoplasia in the head and neck region
* patients affected by gross craniofacial deformities
* pregnant women
* previous UA surgery for OSA
* patients undergoing any other treatment for OSA.

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The patients were recruited in a center for the treatment of obesity after being referenced by the general practitioner to bariatric surgery. All patients apt for the bariatric surgery have attended weekly multi-professional accompaniment (medical, nursing, nutritional, physiotherapy and psychology) for a 16-week period, being subjected to weight loss through diet counselling, practice of physical activities and changes in life habits. The clinical and polysomnographic evaluations for this study have been carried out between 1 and 7 days before the bariatric surgeries. The magnetic resonance of the upper airways was performed on the eve of the bariatric surgery. At least 6 months after the surgeries, patients underwent a repeated polysomnography and Magnetic Resonance.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Upper airway changes after surgical weight loss | 6 months
  Changes in weight (kilograms) measured before and six months after the bariatric surgery.
Obstructive sleep apnea parameters measured thought polysomnographic changes after weight loss | 6 months
  Comparison of pre and post polysomnographic indexes: (apnea hypopnea index (AHI), arousals index, AHI at rapid eye movement (REM) sleep, AHI at supine position)
Changes in volumes and areas of upper airway | 6 months
  Changes through MRI of measures upper airway and volume of tissues, as the percent of fat tissue within (in millimeters and %)
Correlation between the changes on upper airway with the changes on obstructive sleep apnea | 6 months
  Pearson correlation between the changes occurred on upper airway measures and polysomnographic after the procedure

SECONDARY OUTCOMES:
Evaluation if the menstrual status interfere on outcomes | 6 months
  Participants are divided between menses and menopause groups; evaluation of the changes occurred on weight (kilograms), upper airway measures (millimeters and percentages) and polysomnographic (apnea hypopnea indexes) are different according menstrual status

CONTACTS AND LOCATIONS:
Overall Officials: Michel Cahali, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Fundação Hospitalar São Lucas, Cascavel, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
as described in the informed consent form, the data collected in the research would not be shared with the patients, but they could, at the end of the study, request copies of the tests performed.